CLINICAL TRIAL: NCT00761319
Title: An Evaluation of the Ocular Surface Health in Subjects Using TRAVATAN Z® Ophthalmic Solution Versus XALATAN® Ophthalmic Solution
Brief Title: Phase III Clinical Trial of TRAVATAN Z in Ocular Surface Health
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-08-047
Record Dates: First submitted 2008-09-25; First posted 2008-09-29 (Estimated); Results first posted 2012-04-23 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2012-04

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
Keywords: Open-angle glaucoma; ocular hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Travoprost; Latanoprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Travoprost (Experimental): One drop self-administered in the study eye(s) once daily for 90 days
  Interventions: Drug: Travoprost ophthalmic solution 0.004% with SofZia® preservative system (TRAVATAN Z®)
- Latanoprost (Active Comparator): One drop self-administered in the study eye(s) once daily for 90 days
  Interventions: Drug: Latanoprost ophthalmic solution 0.005% (XALATAN®)

INTERVENTIONS:
Drug: Travoprost ophthalmic solution 0.004% with SofZia® preservative system (TRAVATAN Z®) — Ophthalmic solution for the treatment of open-angle glaucoma or ocular hypertension, one drop a day, dosed topically for 90 days. Referred to as travoprost.
  Other Names: TRAVATAN Z®
  Arms: Travoprost
Drug: Latanoprost ophthalmic solution 0.005% (XALATAN®) — Ophthalmic solution for the treatment of open-angle glaucoma or ocular hypertension, one drop a day, dosed topically for 90 days. Referred to as latanoprost.
  Other Names: XALATAN®
  Arms: Latanoprost

SUMMARY:
The purpose of the study is to compare two ophthalmic solutions in patients with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Ocular Surface Disease Index (OSDI) score and corneal fluorescein staining score as specified in protocol.
* Diagnosis of open-angle glaucoma or ocular hypertension in at least one eye.
* Intraocular pressure (IOP) controlled with latanoprost 0.005% (XALATAN®) for at least one continuous month prior to Visit 1.
* Willing and able to discontinue use of any topical ocular medicine other than the study medication for the duration of the study, including artificial tears.
* Best corrected visual acuity of -0.6 logMAR or better in each eye.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any medical condition (systemic or ophthalmic) that may preclude safe administration of the test article.
* Use of contact lenses within 30 days of Visit 1.
* Use of contact lenses during the study.
* Participation in an investigational drug or device study within 30 days of entering this study.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 705 (Actual)
Dates: Start 2008-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 78 US study centers. Eligible patients having a diagnosis of open-angle glaucoma or ocular hypertension and on XALATAN® monotherapy for at least one month immediately prior to Visit 1 were enrolled.
Pre-assignment Details: 705 patients were enrolled in this study. 701 patients were evaluated for safety. Baseline characteristics are presented for all patients who received test article and had at least one on-therapy visit (intent to treat): 652.
Period: Overall Study
Arm/Group | Travoprost | Latanoprost
Started | 353 | 352
Completed | 305 | 318
Not Completed | 48 | 34
Not completed — Protocol Violation | 21 | 14
Not completed — Adverse Event | 11 | 7
Not completed — Withdrawal by Subject | 8 | 7
Not completed — Noncompliance | 4 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Nonspecified | 2 | 2
Not completed — Missing | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Travoprost | Latanoprost | Total
Number analyzed (Participants) | 318 | 334 | 652
Age Continuous [Mean (Standard Deviation); unit: years] | 66.3 (11.8) | 66.3 (10.9) | 66.3 (11.4)
Gender [Number; unit: participants] — One gender response is missing from the Travatan Z arm.
  participants
    Female | 185 | 216 | 401
    Male | 132 | 118 | 250

OUTCOME MEASURES:

1. Primary Outcome: Mean Change at Day 90 From Baseline (Day 0) in Ocular Surface Disease Index (OSDI) Score
Description: The OSDI is a 12-question validated questionnaire (resultant overall 0-100 score) used to measure ocular symptoms, visual function, and environmental factors that may affect a patient's vision, where 0 = normal and 100 = severe. The OSDI questionnaire was administered at both visits and completed by the patient with no assistance from the office staff, physician, or anyone else. A negative number represents a perceived improvement in ocular health.
Time Frame: Day 0, Day 90
Population: Intent to treat. All patients who received test article and had at least one on-therapy study visit were evaluable for the intent-to-treat analysis. Last-observation-carried-forward was used to impute values for dropouts and for missing data on a scheduled study visit during the masked treatment period.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Travoprost | Latanoprost
Number analyzed (Participants) | 305 | 314
Units on a scale | -9.1 (1.0) | -10.2 (0.9)

2. Secondary Outcome: Percentage of Patients With Corneal Fluorescein Staining Score = 0
Description: The corneal surface was assessed by the investigator and graded on a scale of 0-3, where 0 = Absent (no staining present) and 3 = Severe (>50% coverage). Percentage of patients with score = 0 at 90 days was calculated by dividing the number of patients with score = 0 by tht total number of patients analyzed.
Time Frame: Day 90
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Travoprost | Latanoprost
Number analyzed (Participants) | 306 | 318
Percentage of patients | 37.6 | 38.7

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study: 22 October 2008 to 15 September 2009.
Description: This reporting group includes all patients who received the test article. Two patients experienced more than one adverse event.
Arm/Group | Travoprost | Latanoprost
Serious Adverse Events (participants affected / at risk) | 4/353 | 6/348
Other Adverse Events (participants affected / at risk) | 0/353 | 0/348
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Travoprost (N=353) | Latanoprost (N=348)
Cardiac arrest (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
Adverse drug reaction (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Mastectomy (Surgical and medical procedures) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The subjective nature of the OSDI may not be sensitive enough to detect the effects of preservatives on the corneal surface. The measurement and quantification of OSD remains a considerable clinical challenge. (Pflugfelder and Baudoin, 2011)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Alcon reserves the right of prior review of any publication or presentation of information related to the study.